CLINICAL TRIAL: NCT02294123
Title: Glycemic Index and Insulinemic Index of 3 Types of Tortilla in Mexican Adults With Overweight or Diabetes or Clinically Healthy
Brief Title: Glycemic Index and Insulinemic Index of 3 Types of Tortilla in Mexican Adults
Acronym: IGIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Simon Barquera, MD, MS, PhD, Director of Policies and Programs in Nutrition, Mexican National Institute of Public Health
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 120-6526
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes; Overweight; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diabetes (3 tortillas and white bread) (Experimental): Each participants (n=27) receive in random order the following foods: 1) a whole corn tortilla (white "criollo" corn= 5.3% fiber), 2) a whole corn tortilla (white "hybrid" corn= 7.9%), 3) a traditional corn tortilla (3.9% fiber), and 4) white bread (reference food containing 2.2% of fiber).
  Interventions: Other: 3 tortillas and white bread
- Overweight (3 tortillas and white bread) (Experimental): Each participants (n=27) receive in random order the following foods: 1) a whole corn tortilla (white "criollo" corn= 5.3% fiber), 2) a whole corn tortilla (white "hybrid" corn= 7.9%), 3) a traditional corn tortilla (3.9% fiber), and 4) white bread (reference food containing 2.2% of fiber).
  Interventions: Other: 3 tortillas and white bread
- Healthy (3 tortillas and white bread) (Experimental): Each participants (n=27) receive in random order the following foods: 1) a whole corn tortilla (white "criollo" corn= 5.3% fiber), 2) a whole corn tortilla (white "hybrid" corn= 7.9%), 3) a traditional corn tortilla (3.9% fiber), and 4) white bread (reference food containing 2.2% of fiber).
  Interventions: Other: 3 tortillas and white bread

INTERVENTIONS:
Other: 3 tortillas and white bread — Type crossover clinical trial in adults 20-69 years. Three groups of participants were included for each category (n = 27 in each group): 1) adults with diabetes, b) adults with overweight c) clinically healthy adults. The glycemic and insulinemic index was measured for each group of participants given in random order the 3 types of Tortilla and white bread
  Other Names: Glicemic index and insulinemic index

SUMMARY:
Objective. To evaluate the effect of the intake of two types of whole corn tortilla and one traditional tortilla on glycemic index (GI) and insulinemic index (InIn) in adults with diabetes, or overweight or clinically healthy.

Material and methods. Type crossover clinical trial in adults 20-69 years. Three groups of participants will be included for each category (n = 27 in each group): 1) adults with diabetes, b) adults with overweight c) clinically healthy adults. The glycemic and insulinemic index will be measure for each group of participants given in random order the following foods: 1) a whole corn tortilla (white "criollo" corn= 5.3% fiber), 2) a whole corn tortilla (white "hybrid" corn= 7.9%), 3) a traditional corn tortilla (3.9% fiber), and 4) white bread (reference food containing 2.2% of fiber). For the calculation of GI and InIn will be follow the "FAO" methodology. For the evaluation of each food left the range of 1 week.

DETAILED DESCRIPTION:
Objective. To evaluate the effect of the intake of two types of whole corn tortilla, and one traditional tortilla on Glycemic Index (GI) and Insulinemic Index (InIn) in adults with diabetes, or overweight or clinically healthy.

Material and methods. A randomised crossover, single-blinded study design will be undertake in adults 20-69 years. The study will use 3-arm: 1) Adults with diabetes (n=27); b) adults with overweight (n=27); and c) clinically healthy adults (n=27). During a week run-in period subjects will record their normal habitual diet for 7d. Individuals will be request to maintain their normal exercise, and sleeping patterns before reporting for testing.

Upon arrival to the laboratory, participants will be weight and body composition was determined. Overnight fasted (8-12 hours) participants reported to the Research Center of Mexican National Institute of Public Health on 4 occasions separated by at least one week. The glycemic and insulinemic index will be measure for each group of participants given in random order the following foods with a 1-week washout period in between: 1) a whole corn tortilla (white "criollo" corn= 5.3% fiber), 2) a whole corn tortilla (white "hybrid" corn= 7.9%), 3) a traditional corn tortilla (3.9% fiber), and 4) white bread (reference food containing 2.2% of fiber). The rations shall be 50g of carbohydrates available each (approximately equivalent to 4 tortillas or 4 breads, respectively).

Blood samples were collected again at 0, 15, 30, 45, 60, 90 and 120 minutes after completion of the test meal. Insulin and glucose will be measure by electrochemiluminescence and the hexokinase method, respectively. The GI values were determined according to Food and Agriculture Organization of the United Nations (FAO). The area under the curve will be calculated as the incremental area under the blood glucose response curve for each test in each individual. This study and the sampling of the volunteers were performed following approval of the ethics Committee of Mexican National Public Health Institute

ELIGIBILITY:
Inclusion Criteria:

* One group (n=27) with a diagnosis of type 2 diabetes documented by fasting blood glucose.
* One group (n=27) with overweight by Body Mass Index (BMI) >=25 kg/m2
* One group (n=27) with healthy adults without non communicable chronic diseases

Exclusion Criteria:

* Alterations associated with digestion and bariatric surgery

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 2 hours
  Blood glucose concentration increase after food intakes (3 types of tortilla and white bread)
Insulinemic index | 2 hours
  Blood insulin concentration increase after food intakes (3 types of tortilla and white bread)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Barquera, PhD, Principal Investigator — Mexican Institute of Public Health
Locations (1):
- Mexican National Institute of Public Health, Cuernavaca, Morelos, Mexico